CLINICAL TRIAL: NCT00443235
Title: A National, Open-Label, Multicenter, Randomized, Comparative Phase III Study of Induction Treatment With Melphalan/Prednisone/Velcade Versus Thalidomide / Prednisone / Velcade and Maintenance Treatment With Thalidomide / Velcade Versus Prednisone / Velcade in Untreated Patients With Multiple Myeloma More Than 65 Years Old.
Brief Title: GEM05 for Patients With Multiple Myeloma More Than 65 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: pethema, pethema
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-001111-21
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Multiple Myeloma
Keywords: Older patients; untreated patients
MeSH Terms: conditions — Multiple Myeloma | interventions — VMP regimen; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): One cycle:
  Melfalan, 9 mg/m2 v.o days 1 to 4 Prednisone, 60 mg/m2 v.o days 1 to 4 Velcade, 1,3 mg/m2 iv (days 1, 4, 8, 11, 22, 25, 29 and 32) Five cycles: Melfalán, 9 mg/m2 vo, days 1 to 4 Prednisone, 60 mg/m2 v.o days 1 to 4, Velcade,1,3 mg/ m2 iv (days 1, 8, 15 and 22)
  Interventions: Drug: Melphalan/Prednisone/Velcade
- B (Experimental): One cycle:
  Thalidomide,day 1 cycle 1 v.o (50 mg). If toxicity < grade 2, dose will be increased to 100 mg on day 15 cycle 1 Prednisona, 60 mg/m2 vo, days 1 to 4, Velcade, 1,3 mg/ m2 iv (days 1, 4, 8, 11, 22, 25, 29 and 32)
  Five cycles:
  Thalidomide, 100 mg vo all days, Prednisone, 60 mg/m2 vo days 1 to 4, Velcade, 1,3 mg/ m2 iv (days 1, 8, 15 and 22)
  Interventions: Drug: Thalidomide/Prednisone/Velcade

INTERVENTIONS:
Drug: Melphalan/Prednisone/Velcade — One cycle:
  Melfalan, 9 mg/m2 v.o days 1 to 4 Prednisone, 60 mg/m2 v.o days 1 to 4 Velcade, 1,3 mg/m2 iv (days 1, 4, 8, 11, 22, 25, 29 and 32) Five cycles: Melfalán, 9 mg/m2 vo, days 1 to 4 Prednisone, 60 mg/m2 v.o days 1 to 4, Velcade,1,3 mg/ m2 iv (days 1, 8, 15 and 22)
  Arms: A
Drug: Thalidomide/Prednisone/Velcade — One cycle:
  Thalidomide,day 1 cycle 1 v.o (50 mg). If toxicity < grade 2, dose will be increased to 100 mg on day 15 cycle 1 Prednisona, 60 mg/m2 vo, days 1 to 4, Velcade, 1,3 mg/ m2 iv (days 1, 4, 8, 11, 22, 25, 29 and 32)
  Five cycles:
  Thalidomide, 100 mg vo all days, Prednisone, 60 mg/m2 vo days 1 to 4, Velcade, 1,3 mg/ m2 iv (days 1, 8, 15 and 22)
  Arms: B

SUMMARY:
The primary objective is to analyze and compare the efficacy, the response rate, the CR and the response rate duration of both induction treatments and both maintenance treatments

DETAILED DESCRIPTION:
A total of up to 260 patients > 65 years old diagnosed of Multiple Myeloma with symptomatic disease and that have not received previous chemotherapy for MM will be included.

Patients will be evaluated at scheduled visits in up to three study periods: Pre-treatment, Treatment and Follow up.

The Pre-treatment includes Screening and baseline visits. After providing informed consent, patients will be evaluated for study eligibility and then Patients will be randomized one to one to receive Melphalan+Prednisone+Velcade (Group A) or Thalidomide+Prednisone+Velcade (Group B). All of them will received the induction treatment up to 30 weeks. After 4 weeks, without progression and unacceptable toxicity, Patients will be again randomized one to one to receive maintenance treatment: Thalidomide+Velcade (Group M1) or Prednisone+Velcade (Group M2) during three years.

Once the treatment period has finished a follow up will be carry out. During this period we will evaluated response, progression-free survival and global survival every three months.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to comply with the protocol requirements.
* Must voluntary sign the informed consent before performance of any study-related procedure not part of normal medical care, with the understanding it can be withdrawn at any time without prejudice to future medical care.
* Age > 65 years.
* Patient recently diagnosed with symptomatic Multiple Myeloma based on standard criteria28 and that has not received any previous chemotherapy treatment for Multiple Myeloma Some steroid doses or bisphosphonates are allowed for emergencies before starting induction treatment.
* Patient has measurable disease, defined as follows:

For secretory multiple myeloma, measurable disease is defined as any quantifiable serum monoclonal protein value and, where applicable, urine light-chain excretion of ≥ 200 mg/24 hours.

* Patient has a ECOG performance status < 2
* Patient has a life-expectancy >3 months.
* Patient has the following laboratory values before beginning induction treatment:

Platelet count ≥ 50000/mm3, hemoglobin ≥ 8 g/dl and absolute neutrophil count ≥ 1000/mm3. Lower values are allowed if they are due to marrow infiltration.

Corrected serum calcium <14mg/dl. Aspartate transaminase (AST): ≤ 2.5 x the upper limit of normal. Alanine transaminase (ALT): ): ≤ 2.5 x the upper limit of normal. Total bilirubin: ≤1.5 x the upper limit of normal. Serum creatinine ≤ 2 mg/dl.

Exclusion Criteria:

* Patients previously received treatment to Multiple Myeloma, except steroids doses for urgency or bisphosphonates.
* Non-secretor Myeloma
* Patients with < Grade 2 peripheral neuropathy within 14 days before enrolment.
* Patient had major surgery within 4 weeks before enrolment.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Patient has received other investigational drugs within 30 days before enrolment.
* Patient is known to be seropositive for the human immunodeficiency virus (HIV), Hepatitis B surface antigen-positive or active hepatitis C infection.
* Patient had a myocardial infarction within 6 months of enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Patient is enrolled in another clinical research study and/or is receiving an investigational agent for any reason.

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2005-03; Primary Completion 2007-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary objective is to analyze and compare the efficacy, the response rate, the CR and the response rate duration of both induction treatments and both maintenance treatments | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lahuerta Juan josé, Dr, Principal Investigator — Hospital 12 de Octubre
Locations (77):
- Spain (77):
  - Hospital Royo Villanova, Zaragoza, Aragon
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Fundación Hospital Alcorcón, Alcorcón
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Hospital Regional Universitario Infanta Cristina, Badajoz
  - Hospital de Badalona Germans Trias i Pujol, Badalona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Vall D'Hebron, Barcelona
  - Hospital de Basurto, Basurto
  - Hospital de Cruces, Bilbao
  - Hospital General de Castellón, Castellon
  - Hospital Virgen del Puerto, Cáceres
  - Hospital Nuestra Señora de Alarcos, Ciudad Real
  - Hospital Virgen de la Luz, Cuenca
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital General de Elda, Elda
  - Hospital Universitario de Getafe, Getafe
  - Institut Català d'Oncologia,, Girona
  - Hospital General de Guadalajara, Guadalajara
  - Hospital de San Jorge, Huesca
  - Hospital General de Lanzarote, Lanzarote
  - Complejo Hospitalario Xeral-Calde, Lugo
  - Clínica Moncloa, Madrid
  - Clínica Puerta de Hierro, Madrid
  - Clínica Rúber, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Central de la Defensa, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Doce de Octubre, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Althaia, Xarxa Asistencial de Manresa, Manresa
  - Fundación Hospital Sant Joan de Déu de Martorell, Martorell
  - Hospital de Mérida, Mérida
  - Hospital de Móstoles, Móstoles
  - Hospital General Morales Meseguer, Murcia
  - Hospital Santa María del Rosell, Murcia
  - Hospital Virgen del Castillo de Yecla, Murcia
  - Hospital de Gran Canaria Doctor Negrín, Palma de Gran Canaria
  - Complejo Asistencial Son Dureta, Palma de Mallorca
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Verge del Toro, Palma de Mallorca
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital de Navarra, Pamplona
  - Hospital Virgen del Camino, Pamplona
  - Complejo Hospitalario de Pontevedra_Hospital Montecelo, Pontevedra
  - Complejo Hospitalario de Pontevedra_Hospital Provincial, Pontevedra
  - Corporació Sanitaria Parc Taulí, Sabadell
  - Hospital de Sagunto, Sagunto
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital San Pedro de Alcántara, San Pedro
  - Clínica Sant Camil, Sant Pere de Ribes
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital General de Segovia, Segovia
  - Hospital Joan XXIII, Tarragona
  - Hospital Nuestra Señora del Prado, Toledo
  - Hospital Virgen de la Salud, Toledo
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Francesc de Borja, Valencia
  - Hospital General Básico de la Defensa, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Comarcal Pius de Valls, Valls
  - Complejo Hospitalario Universitario de Vigo, Vigo
  - Comarcal de Vinaros, Vinaròs
  - Hospital Txagorritxu, Vitoria-Gasteiz
  - Hospital de Galdakao, Vizcaya
  - Hospital Virgen de la Concha, Zamora
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- [Background] Greenlee RT, Murray T, Bolden S, Wingo PA. Cancer statistics, 2000. CA Cancer J Clin. 2000 Jan-Feb;50(1):7-33. doi: 10.3322/canjclin.50.1.7. PMID 10735013
- [Background] 2. Longo D. Plasma cell disorders. In : Fauce A, et al. Ed. Harrison's Principles of Internal Medicine. 14th Ed. New York, New York: Mc Graw-Hill; 1998: 712-718.
- [Background] Raje N, Anderson K. Thalidomide--a revival story. N Engl J Med. 1999 Nov 18;341(21):1606-9. doi: 10.1056/NEJM199911183412110. No abstract available. PMID 10564693
- [Background] Holland JR, Hosley H, Scharlau C, Carbone PP, Frei E 3rd, Brindley CO, Hall TC, Shnider BI, Gold GL, Lasagna L, Owens AH Jr, Miller SP. A controlled trial of urethane treatment in multiple myeloma. Blood. 1966 Mar;27(3):328-42. No abstract available. PMID 5933438
- [Background] Alexanian R, Haut A, Khan AU, Lane M, McKelvey EM, Migliore PJ, Stuckey WJ Jr, Wilson HE. Treatment for multiple myeloma. Combination chemotherapy with different melphalan dose regimens. JAMA. 1969 Jun 2;208(9):1680-5. doi: 10.1001/jama.208.9.1680. No abstract available. PMID 5818682
- [Background] Salmon SE, Haut A, Bonnet JD, Amare M, Weick JK, Durie BG, Dixon DO. Alternating combination chemotherapy and levamisole improves survival in multiple myeloma: a Southwest Oncology Group Study. J Clin Oncol. 1983 Aug;1(8):453-61. doi: 10.1200/JCO.1983.1.8.453. PMID 6366141
- [Background] Boccadoro M, Marmont F, Tribalto M, Avvisati G, Andriani A, Barbui T, Cantonetti M, Carotenuto M, Comotti B, Dammacco F, et al. Multiple myeloma: VMCP/VBAP alternating combination chemotherapy is not superior to melphalan and prednisone even in high-risk patients. J Clin Oncol. 1991 Mar;9(3):444-8. doi: 10.1200/JCO.1991.9.3.444. PMID 1999714
- [Background] MacLennan IC, Chapman C, Dunn J, Kelly K. Combined chemotherapy with ABCM versus melphalan for treatment of myelomatosis. The Medical Research Council Working Party for Leukaemia in Adults. Lancet. 1992 Jan 25;339(8787):200-5. doi: 10.1016/0140-6736(92)90004-m. PMID 1346171
- [Background] Oken MM, Harrington DP, Abramson N, Kyle RA, Knospe W, Glick JH. Comparison of melphalan and prednisone with vincristine, carmustine, melphalan, cyclophosphamide, and prednisone in the treatment of multiple myeloma: results of Eastern Cooperative Oncology Group Study E2479. Cancer. 1997 Apr 15;79(8):1561-7. PMID 9118039
- [Background] Blade J, San Miguel JF, Alcala A, Maldonado J, Sanz MA, Garcia-Conde J, Moro MJ, Alonso C, Besalduch J, Zubizarreta A, et al. Alternating combination VCMP/VBAP chemotherapy versus melphalan/prednisone in the treatment of multiple myeloma: a randomized multicentric study of 487 patients. J Clin Oncol. 1993 Jun;11(6):1165-71. doi: 10.1200/JCO.1993.11.6.1165. PMID 8501503
- [Background] Combination chemotherapy versus melphalan plus prednisone as treatment for multiple myeloma: an overview of 6,633 patients from 27 randomized trials. Myeloma Trialists' Collaborative Group. J Clin Oncol. 1998 Dec;16(12):3832-42. doi: 10.1200/JCO.1998.16.12.3832. PMID 9850028
- [Background] Richardson PG, Barlogie B, Berenson J, Singhal S, Jagannath S, Irwin D, Rajkumar SV, Srkalovic G, Alsina M, Alexanian R, Siegel D, Orlowski RZ, Kuter D, Limentani SA, Lee S, Hideshima T, Esseltine DL, Kauffman M, Adams J, Schenkein DP, Anderson KC. A phase 2 study of bortezomib in relapsed, refractory myeloma. N Engl J Med. 2003 Jun 26;348(26):2609-17. doi: 10.1056/NEJMoa030288. PMID 12826635
- [Background] Jagannath S, Barlogie B, Berenson J, Siegel D, Irwin D, Richardson PG, Niesvizky R, Alexanian R, Limentani SA, Alsina M, Adams J, Kauffman M, Esseltine DL, Schenkein DP, Anderson KC. A phase 2 study of two doses of bortezomib in relapsed or refractory myeloma. Br J Haematol. 2004 Oct;127(2):165-72. doi: 10.1111/j.1365-2141.2004.05188.x. PMID 15461622
- [Background] 14. Paul Richardson et al. Bortezomib Demonstrates Superior Efficacy to High-Dose Dexamethasone in Relapsed Multiple Myeloma: Final Report of the APEX Study. Blood 2004; 104(11):Abstract number 336.5
- [Background] Rajkumar SV, Hayman S, Gertz MA, Dispenzieri A, Lacy MQ, Greipp PR, Geyer S, Iturria N, Fonseca R, Lust JA, Kyle RA, Witzig TE. Combination therapy with thalidomide plus dexamethasone for newly diagnosed myeloma. J Clin Oncol. 2002 Nov 1;20(21):4319-23. doi: 10.1200/JCO.2002.02.116. PMID 12409330
- [Background] Weber D, Rankin K, Gavino M, Delasalle K, Alexanian R. Thalidomide alone or with dexamethasone for previously untreated multiple myeloma. J Clin Oncol. 2003 Jan 1;21(1):16-9. doi: 10.1200/JCO.2003.03.139. PMID 12506164
- [Background] Rajkumar SV. Thalidomide in newly diagnosed multiple myeloma and overview of experience in smoldering/indolent disease. Semin Hematol. 2003 Oct;40(4 Suppl 4):17-22. doi: 10.1053/j.seminhematol.2003.09.007. PMID 15015892
- [Background] 18. Antonio Palumbo, Alessandra Bertola, Pellegrino Musto, Tommaso Caravita, Vincenzo Callea, Clotilde Cangialosi, Anna Marina Liberati, Pasquale Niscola, Lucio Catalano, Mariella Grasso, Vito Michele Lauta, Maria Concetta Petti, Sergio Morandi, Monica Galli, Sara Bringhen, Federica Cavallo, Patrizia Falco, Mario Boccadoro. A Prospective Randomized Trial of Oral Melphalan, Prednisone, Thalidomide (MPT) vs Oral Melphalan, Prednisone (MP): An Interim Analysis. Blood 2004. Volume 104, issue 11.Abstract number 207
- [Background] 19. Maurizio Zangari, Bart Barlogie, Joth Jacobson, Erik Rasmussen, Michael Burns, Bob Kordsmeier, John D. Shaughnessy, Elias J. Anaissie, Raymond Thertulien, Athanasios Fassas, Choon-Kee Lee, David Schenkein, Jerome B. Zeldis, Guido Tricot. VTD Regimen Comprising Velcade (V) + Thalidomide (T) and Added DEX (D) for Non-Responders to V + T Effects a 57% PR Rate among 56 Patients with Myeloma (M) Relapsing after Autologous Transplant. Blood 2003, Volume 102, issue 11. Abstract number 830
- [Background] 20. Jagannath S, Brian D, Wolf j, Camacho E, Irwin D, Lutzky J, Mckinley M, Gabayan E, Mazumder A, Crowley K, Sckenkein D. A phase 2 study of Bortezomib as first-line therapy in patients with multiple myeloma. Blood 2004; 104(11). Abstract number 333
- [Background] 21. Alexanian R, Wang L, Weber D, Delasalle K. VTD (Velcade, Thalidomide, Dexamethasone) as primary therapy for newly-diagnosed multiple myeloma. Blood 2004; 104(11). Abstract number 210
- [Background] Mateos MV, Hernandez JM, Hernandez MT, Gutierrez NC, Palomera L, Fuertes M, Diaz-Mediavilla J, Lahuerta JJ, de la Rubia J, Terol MJ, Sureda A, Bargay J, Ribas P, de Arriba F, Alegre A, Oriol A, Carrera D, Garcia-Larana J, Garcia-Sanz R, Blade J, Prosper F, Mateo G, Esseltine DL, van de Velde H, San Miguel JF. Bortezomib plus melphalan and prednisone in elderly untreated patients with multiple myeloma: results of a multicenter phase 1/2 study. Blood. 2006 Oct 1;108(7):2165-72. doi: 10.1182/blood-2006-04-019778. Epub 2006 Jun 13. PMID 16772605
- [Background] Whealthy K (On behalf of the Myeloma Trialists'Collaborative Group). Which myeloma patients benefit from interferon therapy?. An overview of 24 randomised trials with 4,000 patients, Br J Haematol 1998; 102: 140
- [Background] Blade J, Esteve J. Viewpoint on the impact of interferon in the treatment of multiple myeloma: benefit for a small proportion of patients? Med Oncol. 2000 May;17(2):77-84. doi: 10.1007/BF02796202. PMID 10871813
- [Background] Palumbo A, Boccadoro M, Garino LA, Gallone G, Frieri R, Pileri A. Multiple myeloma: intensified maintenance therapy with recombinant interferon-alpha-2b plus glucocorticoids. Eur J Haematol. 1992 Aug;49(2):93-7. doi: 10.1111/j.1600-0609.1992.tb00037.x. PMID 1397246
- [Background] Salmon SE, Crowley JJ, Balcerzak SP, Roach RW, Taylor SA, Rivkin SE, Samlowski W. Interferon versus interferon plus prednisone remission maintenance therapy for multiple myeloma: a Southwest Oncology Group Study. J Clin Oncol. 1998 Mar;16(3):890-6. doi: 10.1200/JCO.1998.16.3.890. PMID 9508170
- [Background] Berenson JR, Crowley JJ, Grogan TM, Zangmeister J, Briggs AD, Mills GM, Barlogie B, Salmon SE. Maintenance therapy with alternate-day prednisone improves survival in multiple myeloma patients. Blood. 2002 May 1;99(9):3163-8. doi: 10.1182/blood.v99.9.3163. PMID 11964279
- [Background] International Myeloma Working Group. Criteria for the classification of monoclonal gammopathies, multiple myeloma and related disorders: a report of the International Myeloma Working Group. Br J Haematol. 2003 Jun;121(5):749-57. PMID 12780789
- [Background] Blade J, Samson D, Reece D, Apperley J, Bjorkstrand B, Gahrton G, Gertz M, Giralt S, Jagannath S, Vesole D. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol. 1998 Sep;102(5):1115-23. doi: 10.1046/j.1365-2141.1998.00930.x. No abstract available. PMID 9753033
- [Background] Rizzo JD, Lichtin AE, Woolf SH, Seidenfeld J, Bennett CL, Cella D, Djulbegovic B, Goode MJ, Jakubowski AA, Lee SJ, Miller CB, Rarick MU, Regan DH, Browman GP, Gordon MS; American Society of Clinical Oncology; Americcan Society of Hematology. Use of epoetin in patients with cancer: evidence-based clinical practice guidelines of the American Society of Clinical Oncology and the American Society of Hematology. Blood. 2002 Oct 1;100(7):2303-20. doi: 10.1182/blood-2002-06-1767. PMID 12239138
- [Background] Rizzo JD, Lichtin AE, Woolf SH, Seidenfeld J, Bennett CL, Cella D, Djulbegovic B, Goode MJ, Jakubowski AA, Lee SJ, Miller CB, Rarick MU, Regan DH, Browman GP, Gordon MS; American Society of Clinical Oncology. American Society of Hematology. Use of epoetin in patients with cancer: evidence-based clinical practice guidelines of the American Society of Clinical Oncology and the American Society of Hematology. J Clin Oncol. 2002 Oct 1;20(19):4083-107. doi: 10.1200/JCO.2002.07.177. PMID 12351606
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] 33. Fayers P, Aaonson N, Bjordal K, Curran D, Groenvold M, on behalf of the EORTC Quality of life study group. EORTC QLQ-C30 Scoring Manual: 2nd Ed. 1999. ISBN 2-930064-16-1.1
- [Background] Stead ML, Brown JM, Velikova G, Kaasa S, Wisloff F, Child JA, Hippe E, Hjorth M, Sezer O, Selby P. Development of an EORTC questionnaire module to be used in health-related quality-of-life assessment for patients with multiple myeloma. European Organization for Research and Treatment of Cancer Study Group on Quality of Life. Br J Haematol. 1999 Mar;104(3):605-11. doi: 10.1046/j.1365-2141.1999.01206.x. PMID 10086801
- [Derived] Mateos MV, Oriol A, Martinez-Lopez J, Teruel AI, Bengoechea E, Palomera L, de Arriba F, Esseltine DL, Cakana A, Pei L, van de Velde H, Miguel JS. Outcomes with two different schedules of bortezomib, melphalan, and prednisone (VMP) for previously untreated multiple myeloma: matched pair analysis using long-term follow-up data from the phase 3 VISTA and PETHEMA/GEM05 trials. Ann Hematol. 2016 Dec;95(12):2033-2041. doi: 10.1007/s00277-016-2835-3. Epub 2016 Oct 14. PMID 27738789
- [Derived] Mateos MV, Martinez-Lopez J, Hernandez MT, Ocio EM, Rosinol L, Martinez R, Teruel AI, Gutierrez NC, Martin Ramos ML, Oriol A, Bargay J, Bengoechea E, Gonzalez Y, Perez de Oteyza J, Gironella M, Encinas C, Martin J, Cabrera C, Paiva B, Cedena MT, Puig N, Blade J, Lahuerta JJ, San-Miguel J. Sequential vs alternating administration of VMP and Rd in elderly patients with newly diagnosed MM. Blood. 2016 Jan 28;127(4):420-5. doi: 10.1182/blood-2015-08-666537. Epub 2015 Oct 23. PMID 26500339
- [Derived] Mateos MV, Oriol A, Martinez-Lopez J, Teruel AI, Lopez de la Guia A, Lopez J, Bengoechea E, Perez M, Martinez R, Palomera L, de Arriba F, Gonzalez Y, Hernandez JM, Granell M, Bello JL, Bargay J, Penalver FJ, Martin-Mateos ML, Paiva B, Montalban MA, Blade J, Lahuerta JJ, San-Miguel JF. GEM2005 trial update comparing VMP/VTP as induction in elderly multiple myeloma patients: do we still need alkylators? Blood. 2014 Sep 18;124(12):1887-93. doi: 10.1182/blood-2014-05-573733. PMID 25102853
- [Derived] Martinez-Lopez J, Fernandez-Redondo E, Garcia-Sanz R, Montalban MA, Martinez-Sanchez P, Pavia B, Mateos MV, Rosinol L, Martin M, Ayala R, Martinez R, Blanchard MJ, Alegre A, Besalduch J, Bargay J, Hernandez MT, Sarasquete ME, Sanchez-Godoy P, Fernandez M, Blade J, San Miguel JF, Lahuerta JJ; GEM (Grupo Espanol Multidisciplinar de Melanoma)/PETHEMA (Programa para el Estudio de la Terapeutica en Hemopatias Malignas) cooperative study group. Clinical applicability and prognostic significance of molecular response assessed by fluorescent-PCR of immunoglobulin genes in multiple myeloma. Results from a GEM/PETHEMA study. Br J Haematol. 2013 Dec;163(5):581-9. doi: 10.1111/bjh.12576. Epub 2013 Oct 3. PMID 24117042
- [Derived] Mateos MV, Oriol A, Martinez-Lopez J, Gutierrez N, Teruel AI, Lopez de la Guia A, Lopez J, Bengoechea E, Perez M, Polo M, Palomera L, de Arriba F, Gonzalez Y, Hernandez JM, Granell M, Bello JL, Bargay J, Penalver FJ, Ribera JM, Martin-Mateos ML, Garcia-Sanz R, Lahuerta JJ, Blade J, San-Miguel JF. Maintenance therapy with bortezomib plus thalidomide or bortezomib plus prednisone in elderly multiple myeloma patients included in the GEM2005MAS65 trial. Blood. 2012 Sep 27;120(13):2581-8. doi: 10.1182/blood-2012-05-427815. Epub 2012 Aug 13. PMID 22889759
- [Derived] Lopez-Corral L, Mateos MV, Corchete LA, Sarasquete ME, de la Rubia J, de Arriba F, Lahuerta JJ, Garcia-Sanz R, San Miguel JF, Gutierrez NC. Genomic analysis of high-risk smoldering multiple myeloma. Haematologica. 2012 Sep;97(9):1439-43. doi: 10.3324/haematol.2011.060780. Epub 2012 Feb 13. PMID 22331267
- [Derived] Mateos MV, Gutierrez NC, Martin-Ramos ML, Paiva B, Montalban MA, Oriol A, Martinez-Lopez J, Teruel AI, Bengoechea E, Martin A, Diaz-Mediavilla J, de Arriba F, Palomera L, Hernandez JM, Sureda A, Bargay J, Penalver FJ, Ribera JM, Martin-Mateos ML, Fernandez M, Garcia-Sanz R, Vidriales MB, Blade J, Lahuerta JJ, San Miguel JF. Outcome according to cytogenetic abnormalities and DNA ploidy in myeloma patients receiving short induction with weekly bortezomib followed by maintenance. Blood. 2011 Oct 27;118(17):4547-53. doi: 10.1182/blood-2011-04-345801. Epub 2011 Sep 6. PMID 21900193
- [Derived] Sarasquete ME, Gutierrez NC, Misiewicz-Krzeminska I, Paiva B, Chillon MC, Alcoceba M, Garcia-Sanz R, Hernandez JM, Gonzalez M, San-Miguel JF. Upregulation of Dicer is more frequent in monoclonal gammopathies of undetermined significance than in multiple myeloma patients and is associated with longer survival in symptomatic myeloma patients. Haematologica. 2011 Mar;96(3):468-71. doi: 10.3324/haematol.2010.033845. Epub 2010 Dec 15. PMID 21160068
- [Derived] Mateos MV, Oriol A, Martinez-Lopez J, Gutierrez N, Teruel AI, de Paz R, Garcia-Larana J, Bengoechea E, Martin A, Mediavilla JD, Palomera L, de Arriba F, Gonzalez Y, Hernandez JM, Sureda A, Bello JL, Bargay J, Penalver FJ, Ribera JM, Martin-Mateos ML, Garcia-Sanz R, Cibeira MT, Ramos ML, Vidriales MB, Paiva B, Montalban MA, Lahuerta JJ, Blade J, Miguel JF. Bortezomib, melphalan, and prednisone versus bortezomib, thalidomide, and prednisone as induction therapy followed by maintenance treatment with bortezomib and thalidomide versus bortezomib and prednisone in elderly patients with untreated multiple myeloma: a randomised trial. Lancet Oncol. 2010 Oct;11(10):934-41. doi: 10.1016/S1470-2045(10)70187-X. Epub 2010 Aug 23. PMID 20739218
- See also: Spanish association of Haematology — http://www.aehh.org